CLINICAL TRIAL: NCT07259577
Title: Effects of Vagus Nerve Stimulation on Motor Function, Respiratory Muscle Strength, and Quality of Life in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yusuf AÇIKGÖZ, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1439695
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Stroke Treatment
Keywords: stroke; Upper Extremity Robot-Assisted Training; Transcutaneous Auricular Vagus Nerve Stimulation; taVNS; Respiratory Muscle Strength
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotics Assisted Education + taVNS (Active Comparator)
  Interventions: Device: Robotics Assisted Education + taVNS
- Robotics Assisted Education + sham (Sham Comparator)
  Interventions: Other: Robotics Assisted Education + sham

INTERVENTIONS:
Device: Robotics Assisted Education + taVNS — Conventional rehabilitation will be administered 3 days a week, 45 minutes per day, for 5 weeks. The combination of Upper Extremity Robotic-Assisted Training and Transcutaneous Auricular Vagus Nerve Stimulation will be administered 2 days a week, 45 minutes per day, for 5 weeks.
  Arms: Robotics Assisted Education + taVNS
Other: Robotics Assisted Education + sham — Conventional rehabilitation will be administered 3 days a week, 45 minutes per day, for 5 weeks. The combination of Upper Extremity Robotic-Assisted Training and Sham Transcutaneous Auricular Vagus Nerve Stimulation will be administered 2 days a week, 45 minutes per day, for 5 weeks.
  Arms: Robotics Assisted Education + sham

SUMMARY:
Stroke is one of the leading causes of death and permanent disability worldwide. Loss of upper extremity (UE) function after stroke significantly reduces independence and quality of life. Moreover, weakness in the respiratory muscles negatively affects trunk control and respiratory function, limiting overall functional recovery. In recent years, robot-assisted training (RAT) and non-invasive neuromodulation techniques-particularly transcutaneous auricular vagus nerve stimulation (taVNS)-have emerged as promising approaches to enhance neuroplasticity in stroke rehabilitation.

This study aims to investigate the effects of taVNS combined with robot-assisted training on upper extremity motor function, respiratory muscle strength, and quality of life in individuals with stroke.

This randomized controlled trial will be conducted in collaboration between Istanbul University-Cerrahpaşa and Istanbul Medeniyet University. Thirty individuals aged 18-70 years, with moderate-to-severe upper extremity weakness and a history of stroke of at least six months, will be included. Participants will be randomly assigned to two groups: RAT + taVNS (n=15), RAT + sham taVNS (n=15). Both groups will receive conventional rehabilitation for 45 minutes, three times per week for five weeks. Additionally, each group will undergo 45-minute sessions of RAT twice per week for five weeks, with either active or sham taVNS applied concurrently.

The primary outcome measure will be the Fugl-Meyer Upper Extremity Motor Assessment (FM-UE). Secondary outcomes will include the Stroke Impact Scale (SIS), Maximum Inspiratory Pressure (MIP), Maximum Expiratory Pressure (MEP), and Fatigue Assessment Scale (FAS). Assessments will be conducted at baseline and at the end of the fifth week.

Combining taVNS with robot-assisted upper extremity rehabilitation is expected to result in greater improvements in motor function, respiratory muscle strength, and quality of life compared to robot-assisted rehabilitation alone. This study will provide valuable insights into the synergistic effects of neuromodulation and robotic therapy in stroke rehabilitation and contribute to the growing body of evidence supporting non-invasive, technology-assisted treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-70 years diagnosed with ischemic or hemorrhagic stroke lasting longer than 6 months,
* Moderate to severe upper extremity weakness (20-50 out of 66 on the Fugl-Meyer Upper Extremity Motor Assessment Scale),
* Ability to communicate and understand (Mini Mental State Examination (MMSE) score ≥ 23),
* Upper extremity spasticity of 2 or less on the Modified Ashworth Scale.

Exclusion Criteria:

* Use of any stimulation device, such as a pacemaker or other neurostimulator,
* Presence of a medical or cognitive condition (personality disorder, anxiety, depression, etc.) that would prevent participants from participating in the study,
* Receiving a Botox injection into the affected upper extremity at least 4 weeks prior,
* Severe spasticity in the upper extremity (Modified Ashworth Scale ≥3),
* Presence of dysphagia or aphasia,
* Presence of cardiac problems such as atrial fibrillation, atrial flutter, sick sinus syndrome, or atrioventricular block.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Evaluation (FM-UE) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  We will use the Fugl-Meyer Upper Motor Assessment score, which is the most sensitive for treatment outcomes in stroke patients presenting with unilateral paresis in the post-stroke period. It measures upper extremity use and impairment, measuring shoulder, elbow, forearm, wrist, finger, and reflex movements from proximal to distal, synergistic to extrinsic. The score ranges from 0 to 66 and consists of 33 items. 0-28 indicates severe motor impairment; 29-42 indicates moderate motor impairment; and 43-66 indicates mild motor impairment. Higher scores indicate better performance. The FM-UE consists of one component, each rated on a 3-point ordinal scale (0=not achieved, 1=partially contributed, 2=completely contributed). The minimum clinically meaningful change on the FM-UE for chronic stroke has been determined to be 4.25 to 7.25. Consistent with the literature, we define an improvement of at least 6 points or more as significant.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  The SIS 3.0 assesses function and quality of life based on subjective report in eight clinically important domains. It consists of two parts. The first part is the main scale of the IAS, which assesses multidimensional health-related quality of life (QOL) including strength, hand function, ADL/instrumental ADL, mobility, communication, emotion, memory/thinking, and social participation. It consists of 59 items, and each item is subjectively rated by stroke patients on a 5-point Likert-type scale according to their perceived difficulty with the item in the past week. The score for each domain is converted to a score out of 100, and the average scores for all domains are used to represent stroke patients' multidimensional health-related quality of life. The formula Domain Score = [(Average Item Score -1) / (5 -1) x 100] is used to convert each domain score. SIS 3.0 also includes assessment of post-stroke recovery using a 0-100 visual analog scale (0: no recovery, 100: complete recovery)
Maximum Inspiratory Pressure (MIP) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  This is the pressure measured when the patient tries to breathe as forcefully as possible into their lungs (inspiration). It assesses the strength of the diaphragm and accessory respiratory muscles-in other words, the inspiratory capacity of the respiratory muscles. The measurement is taken through the mouth. A nose clip is applied. After maximum exhalation near the residual volume (RV), the patient tries to breathe in as forcefully as possible for 1-2 seconds. Three repetitions are performed, and the average is calculated. (The higher the pressure value, the greater the muscle strength.)
Maximum Expiratory Pressure (MEP) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  This is the pressure measured during the patient's strongest possible exhalation (expiration). This indicates the strength of the respiratory muscles that assist exhalation, such as the abdominal muscles and internal/external intercostal muscles. The measurement is taken orally. A nose clip is applied. After taking a maximum inspiration (close to TLC), the patient attempts to exhale as forcefully as possible for 1-2 seconds. Three repetitions are performed, and the average is calculated. (The higher the pressure value, the greater the muscle strength.)
Fatigue Assessment Scale(FAS) | Outcome measures will be assessed and recorded at baseline (assessment session) and after intervention (week 5).
  It is a brief and practical self-report instrument developed to measure the severity of fatigue experienced by individuals. It consists of 10 items, and each item is rated subjectively on a 5-point Likert-type scale used to assess overall fatigue level over the past week. The lowest score is 10, and the highest is 50. (≤ 21 points: None/low fatigue, 22-34 points: Moderate fatigue, ≥ 35 points: High fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Açıkgöz, Principal Investigator — Istanbul University - Cerrahpasa; Rüstem Mustafaoğlu, Study Director — Istanbul University-Cerrahpasa Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa Sağlık Bilimleri Fakültesi Büyükçekmece Yerleşkesi, Istanbul, Istanbul, Turkey (Türkiye)